CLINICAL TRIAL: NCT04348006
Title: Assessment of Bortezomib (Alvocade ®) Efficacy and Safety in Newly Diagnosed Multiple Myeloma Patients
Acronym: MM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patients were enrolled in the study
Sponsor: Al-Rasheed University College (Other)
Collaborators: Baghdad Medical City (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AR200103; SEANM (Registry Identifier: Baghdad Hematology Center Ethical committee)
Record Dates: First submitted 2020-04-13; First posted 2020-04-15 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Newly Diagnosed Multiple Myeloma
MeSH Terms: interventions — Bortezomib; Cyclophosphamide; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Induction Therapy (Experimental): Bortezomib will be administered as part of VCD or VRD protocols
  Interventions: Drug: Bortezomib 3.5 MG

INTERVENTIONS:
Drug: Bortezomib 3.5 MG — VCD protocol
  * V, Alvocade®: Day 1, 4, 8, 11 (1.3 mg/m2 SC)
  * C, Cyclophosphamide: 300 mg/m2 IV over 30 min (day 1, 8, 15)
  * D, Dexamethasone oral: 40mg (days 1 to 4)
  VRD protocol:
  * V, Alvocade®: Day 1, 4, 8, 11 (1.3 mg/m2 SC)
  * R, Lenalid® cap 25 mg po (day 1 to 21)
  * D, Dexamethasone oral: 40mg (days 1 to 4)
  Other Names: Cyclophosphamide; Dexamethasone; lenalidomide

SUMMARY:
Bortezomib considered the standard of care for treating multiple myeloma patients, the aim was to assess the safety and efficacy of newly approved drug (Alvocade ®) in Iraq, in newly diagnosed patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosis Multiple myeloma with CRAB (C: hypercalcemia, R: renal impairment, A: anemia, and B: bone lesions)
* Age above 18 years old

Exclusion Criteria:

* Age below 18 years
* Smoldering MM

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-07-30 (Estimated); Study Completion 2021-07-30 (Estimated)

PRIMARY OUTCOMES:
Assessment the safety of Alvocade® therapy | During 6 months
  Monitoring the rate of any adverse effect/event that will occur during the induction therapy
Assessment the effecacy of Alvocade® therapy | At end of 6 months
  Assessment of overall response rate (ORR) of treatment after completion of induction protocol

SECONDARY OUTCOMES:
First assessment response | At end of 2 months
  Assessment of response rate after 2 cycle from starting treatment protocol
Second assessment response | At end of 4 months
  Assessment of response rate after 4 cycle from starting treatment protocol
Third assessment response | At end of 6 months
  Third assessment response after 6th cycle protocol (if there is no response or get less than VGPR after 4th cycle)

CONTACTS AND LOCATIONS:
Overall Officials: Ali M Jawad, PhD, Principal Investigator — University of Baghdad; Bassam F Matti, PhD, Principal Investigator — Baghdad Medical City; Tareq A Saleh, PhD, Study Chair — Baghdad Medical City; Mahammed S Abbas, PhD, Study Director — Baghdad Medical City; Mohammed K Al-Qayyim, PhD, Principal Investigator — Baghdad Medical City; Alaaldin S Naji, PhD, Principal Investigator — University of Baghdad; Ammer F Majid, PhD, Principal Investigator — Baghdad Medical City; Adil S Al-Oqaby, PhD, Principal Investigator — Baghdad Medical City; Mazin A Shubir, PhD, Principal Investigator — Baghdad Medical City; Hawraa D Jumaa, PhD, Principal Investigator — Baghdad Medical City; Hayder A Fawzi, PhD, Principal Investigator — Al-Rasheed University College
Locations (1):
- Baghdad Hematology center - Baghdad Medical City, Baghdad, Bab-Almuadham, Iraq

IPD SHARING:
Plan to Share IPD: Undecided